CLINICAL TRIAL: NCT06889558
Title: Evaluation of the Bone Volume in Horizontal Atrophic Ridges Augmentation Using Tenting Grafting Technique Versus Khoury Technique in Mandibular Molar and Premolar Region: Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ABDULRAHMAN RAJAB KHALLEEFAH, Evaluation of the bone volume in Horizontal Atrophic Ridges Augmentation Using Tenting Grafting Technique versus Khoury Technique in mandibular molar and premolar region: Randomized Clinical Trial., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dental Tenting Graft technique
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Augmentation, Alveolar Ridge

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Khoury technique (Active Comparator): technique use for bone augmentation in atrophic ridges
  Interventions: Procedure: tenting titanium screw
- tenting technique (Experimental): technique used for increase bone volume
  Interventions: Procedure: tenting titanium technique

INTERVENTIONS:
Procedure: tenting titanium technique — technique used to increase bone augmentation and increase bone volume
  Other Names: tenting screw
  Arms: tenting technique
Procedure: tenting titanium screw — technique used for increase bone voliume
  Arms: Khoury technique

SUMMARY:
The aim of this study is to compare the effectiveness of the Tenting Grafting Technique and the Khoury Technique for horizontal augmentation of atrophic alveolar ridges in mandibular molar and premolar regions in dental implant procedures.

Hypothesis:

We hypothesis that the tenting grafting technique is more effective for augmenting atrophic ridges with horizontal bone deficiency, whereas the Khoury technique will yield superior results for severely atrophic ridges, where both vertical and horizontal bone augmentation is required.

DETAILED DESCRIPTION:
II. Introduction:

6. Background and rationale:

Research question:

Would the tenting grafting technique result better in horizontal bone augmentation outcomes compared to the Khoury technique for atrophic ridges in dental implant procedures?

Statement of the problem:

Bone augmentation techniques are required in order to improve esthetic outcomes and long-term prognoses for dental implant treatment. These techniques involve the use of bone graft materials for the rehabilitation of deficient regions (Goudarzimoghaddam et al., 2024).

Atrophic ridges, which result from significant bone loss due to tooth extraction or long-term edentulism. The lack of sufficient bone volume can compromise the ability to place dental implants successfully, leading to poor functional and aesthetic outcomes.

However, there is a lack of consensus on which technique provides superior results in terms of bone regeneration, implant stability, complication rates, and overall patient satisfaction. Furthermore, the healing time, risk of complications, and long-term success of these techniques remain subjects of debate.

Rationale for conducting the research:

Tooth loss is accompanied by a series of adaptive changes, leading to dimensional alterations of the alveolar process. During the first year after tooth extraction, Schropp et al. described 50% bone loss in the buccal-lingual dimension, with 30% of the initial ridge width lost during the first 3 months (Hares et al., 2021).

Atrophic ridges present significant challenges in dental implantology, particularly when there is insufficient bone volume for the proper placement of implants. Ridge augmentation techniques become essential to restore the lost bone and ensure a stable foundation for implants (Goudarzimoghaddam et al., 2024). Bone augmentation techniques are required in order to improve esthetic outcomes and long-term prognoses for dental implant treatment. These techniques involve the use of bone graft materials for the rehabilitation of deficient regions (Işık et al., 2021).

Bone graft materials originating from human, animal, or synthetic sources are placed to induce osteoblastic activity of the bone and periosteal tissue, or to provide an osteoconductive scaffold that indirectly accelerates bone regeneration. These materials are manufactured in block or particulate forms to allow them to adapt to different bone defects (César Neto et al., 2020).

While the block forms have good mechanical properties, the particulate forms can have some disadvantages in reconstructing alveolar bone deficiencies, namely soft tissue migration, lack of structural integrity, which affects stability and also the collapse of the bone graft materials. Two of the commonly used methods for augmenting atrophic ridges are the tenting grafting technique and the Khoury technique (Abo Zekry et al., 2024) .

In the last decade, "tent-pole" techniques have been introduced to prevent the contraction of soft tissue around the bone graft material and to reduce micromovement or physiological resorption of the grafts. These techniques are a relatively newer and innovative method, create a space between the bone and periosteum for particulate grafts and provide ample bone volume. It is primarily used for horizontal bone augmentation, particularly in cases where the ridge is severely resorbed, making it difficult to place implants without bone grafting. This technique involves the use of a tenting screw or titanium mesh, which acts as a "tent" to support the bone graft material and prevent its collapse (Hares et al., 2021).

Within the wide range of different augmentation procedures, guided bone regeneration (GBR) and the use of autogenous bone blocks are the most common interventions in bone augmentation; Khoury et al. is a well-established method for augmenting atrophic bone ridges, described the stabilization of two split autologous bone blocks by microscrews and filling the generated gap with autogenous bone chips. These split bone blocks are obtained, either from the mandibular symphysis or ramus, using piezoelectric surgery or microsaws, obtaining a block that will later be divided into the two final thin laminae (Urban et al., 2023).

However, there is a lack of consensus on which technique provides superior results in terms of bone regeneration, implant stability, complication rates, and overall patient satisfaction. Hence, this study aims to evaluate atrophic ridges augmentation using tenting grafting technique versus Khoury technique.

Explanation for choice of comparators:

Both techniques are commonly employed in clinical practice for augmenting atrophic bone ridges, particularly when there is insufficient bone volume for dental implant placement. Comparing them provides meaningful insights into which method might offer better outcomes for patients with these common challenges.

7. Objectives: The aim of this study is to compare the effectiveness of the Tenting Grafting Technique and the Khoury Technique for horizontal augmentation of atrophic alveolar ridges in dental implant procedures.

Hypothesis:

We hypothesis that the tenting grafting technique is more effective for augmenting atrophic ridges with horizontal bone deficiency, whereas the Khoury technique will yield superior results for severely atrophic ridges, where both vertical and horizontal bone augmentation is required.

8. Trial design:

* Randomized clinical trial.
* Parallel group study.
* Allocation ratio 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Cooperative and likely to maintain good dental health.
* Adequate bone height for placement of implants with a minimum length of 10 mm.
* Totally or partially edentulous alveolar ridges.
* Placement Patients with insufficient bone for an implant.

Exclusion criteria:

* Presence of any local or systemic factors that might contraindicate oral surgery.
* Poor oral hygiene. Conditions that complicate wound healing such as uncontrolled diabetes, smoking (10 cigarettes a day), pregnancy, a history of drug or alcohol abuse, and an inability or unwillingness to return for follow ups after occlusal loading
* Pathological lesions in the defect site.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or para-functional habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain and volume by CBCT | baseline
  measurement of bone volume by CBCT in cubic centimeter ( cc3 )

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Angelis P, Cavalcanti C, Manicone PF, Liguori MG, Rella E, De Rosa G, Palmieri A, D'Addona A. A Comparison of Guided Bone Regeneration vs. the Shell Technique Using Xenogeneic Bone Blocks in Horizontal Bone Defects: A Randomized Clinical Trial. Dent J (Basel). 2024 May 9;12(5):137. doi: 10.3390/dj12050137. PMID 38786535